CLINICAL TRIAL: NCT00204737
Title: A Placebo-controlled, Randomized, Double-blind Comparison of Placebo vs Short Course Low Dose Corticosteroids on Posttraumatic Stress Disorder (PTSD)
Brief Title: Short Course Glucocorticoid Treatment for PTSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-2004-0039
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisone (Active Comparator): Prednisone 20mg daily x 2 weeks
  Interventions: Drug: prednisone
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prednisone — 20mg x 2 weeks
  Arms: Prednisone
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate if a 2-wk course of 20mg/day of oral prednisone in addition to standard care will result in reduced PTSD symptoms or symptom severity compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Must meet Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for PTSD w/ symptom exacerbation (CAPS score ≥ 50)
* Stable on other psychotropic meds x1 month

Exclusion Criteria:

* Current or past history of bipolar, schizophrenic, or other psychotic disorder
* Organic mental disorder
* Alcohol or substance abuse in last 3 months
* Clinically significant hepatic or renal disease or other acute or unstable medical condition
* Chronic obstructive pulmonary disease (COPD), asthma, uncontrolled diabetes, rheumatologic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine D. Johnson, PharmD, MS, BCPP, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Catherine Johnson, Madison, Wisconsin
  - Wm. S. Middleton VA Hospital, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prednisone | Placebo
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (10.3) | 56.0 (4.9) | 54 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Marital Status [Count of Participants; unit: Participants]
  Married | 2 | 2 | 4
  Divorced | 3 | 4 | 7
  Widowed | 1 | 0 | 1
Trauma Type [Count of Participants; unit: Participants]
  Combat | 5 | 4 | 9
  Childhood Abuse | 1 | 1 | 2
  Employment | 0 | 1 | 1
Education Level [Count of Participants; unit: Participants]
  High School / GED | 3 | 4 | 7
  Some College | 1 | 1 | 2
  Bachelor's or Technical School | 2 | 1 | 3
Percent Service Connection [Count of Participants; unit: Participants] — Disability compensation is a monetary benefit paid to Veterans determined by the VA to be disabled by an injury or illness that was incurred or aggravated during active military service.
  Participants
    0 percent | 1 | 1 | 2
    1-30 percent | 0 | 2 | 2
    31-60 percent | 0 | 0 | 0
    61-99 percent | 3 | 3 | 6
    100 percent | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Administered PTSD Scale (CAPS)
Description: This measure tests the hypothesis that there will be a 30% or greater improvement in the Clinician-Administered PTSD (Post Traumatic Stress Disorder) Scale over the course of the study. CAPS is a 30-item survey with a total possible range of scores from 0-120 where the higher the score, the more severe the symptoms.
Time Frame: baseline, 2 weeks, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 96.0 (17.1) | 90.7 (13.3)
  2 Weeks | 66.3 (18.6) | 86.2 (21.0)
  6 Weeks | 72.8 (18.2) | 81.5 (11.6)
  12 Weeks | 75.2 (27.0) | 82.5 (18.7)

2. Primary Outcome: Number of Participants Achieving CAPS Response
Description: CAPS response defined as a 30% reduction in CAPS score from baseline.
Time Frame: baseline, 2 weeks, 6 weeks, 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 6
Participants
  baseline to 2 weeks | 4 | 0
  baseline to 6 weeks | 3 | 0
  baseline to 12 weeks | 1 | 0
Statistical Analysis 1: Comparison: Prednisone vs Placebo; comparison at 2 Weeks; Test type: Other; p = 0.06, Fisher Exact
Statistical Analysis 2: Comparison: Prednisone vs Placebo; Comparison at 6 Weeks; Test type: Other; p = 0.18, Fisher Exact
Statistical Analysis 3: Comparison: Prednisone vs Placebo; Comparison at 12 weeks; Test type: Other; p = 0.5, Fisher Exact

3. Secondary Outcome: Change in Hamilton Depression Rating Scale (HAM-D)
Description: HAM-D is a 21-item survey where scoring is based on the first 17-items. It has a total possible range of scores 0-50 where higher scores indicate more severe depression.
Time Frame: baseline, 2 weeks, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 19.2 (7.2) | 16.8 (5.8)
  2 Weeks | 13.2 (6.1) | 14.8 (6.7)
  6 Weeks | 11.7 (5.9) | 14.5 (6.2)
  12 Weeks | 12.3 (5.7) | 15.7 (5.9)

4. Secondary Outcome: Change in PCL-PTSD Score
Description: PCL-PTSD is a 17-item survey with a total possible range of scores 17-85 where higher scores indicate more severe symptoms.
Time Frame: baseline, 2 weeks, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 68.7 (10.6) | 64.2 (9.5)
  2 Weeks | 58.8 (7.5) | 59.8 (8.0)
  6 Weeks | 56.0 (13.3) | 60.3 (6.0)
  12 Weeks | 58.2 (15.6) | 64.2 (8.4)

5. Secondary Outcome: Change in Clinical Global Impression Severity (CGI-S) Score
Description: CGI-S is scored by a clinician. It is a 7 point scale where 1 = normal, 2 = borderline mentally ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill.
Time Frame: baseline, 2 weeks, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 5.5 (1.0) | 5.5 (0.8)
  2 Weeks | 4.7 (0.8) | 5.5 (0.8)
  6 Weeks | 4.8 (0.8) | 5.2 (0.8)
  12 Weeks | 4.5 (1.0) | 5.5 (1.0)

6. Secondary Outcome: Change in Dehydroepiandrosterone Sulfate (DHEA-S)
Description: DHEA-S measured at baseline, 2 weeks, 6 weeks, and 12 weeks
Time Frame: Baseline, 2 weeks, 6 weeks, and 12 weeks
Measure: Mean (Standard Deviation); unit: mcg/dl
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 6
mcg/dl
  Baseline | 123.8 (115.0) | 201.2 (280.2)
  2 Weeks | 87.7 (105.6) | 148.7 (170.8)
  6 Weeks | 123.5 (116.2) | 156.8 (188.3)
  12 Weeks | 112.3 (117.4) | 157.8 (211.8)

7. Secondary Outcome: Change in Salivary Cortisol (First 6 Participants)
Time Frame: Baseline, 2 weeks, 6 weeks, and 12 weeks
Population: Midway through the study, the protocol related to salivary cortisol was modified to add the dexamethasone suppression test to better understand response of the hypothalamic pituitary adrenal (HPA) axis to a steroid challenge. This is why no participants were analyzed during week 2.
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 3 | 3
ug/dl
  Baseline | 0.13 (0.05) | 0.08 (0.03)
  2 Weeks: number analyzed (Participants) | 0 | 0
  6 Weeks | 0.10 (0.02) | 0.09 (0.03)
  12 Weeks | 0.10 (0.01) | 0.07 (0.03)

8. Secondary Outcome: Change in Salivary Cortisol (Last 6 Participants)
Description: Participants provided saliva samples at 16:00, 24:00, and 08:00. After these samples are collected, participants take 0.5mg dexamethasone orally at 23:00, and a fourth sample is collected at 08:00 post dexamethasone. Post-dexamethasone data is reported here.
Time Frame: Baseline, 2 weeks, 6 weeks, and 12 weeks
Population: One participant in the Prednisone arm did not provide enough sample for analysis and one additional participant in the Prednisone arm did not provide enough sample for analysis at week 6. Data was not collected for week 2 due to protocol amendment to change cortisol testing.
Measure: Mean (Standard Deviation); unit: ug/dl
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 2 | 3
ug/dl
  Baseline | 0.1 (0.1) | 0.138 (0.067)
  2 Weeks: number analyzed (Participants) | 0 | 0
  6 Weeks: number analyzed (Participants) | 1 | 3
  6 Weeks | 0.103 (NA) — Only one data point. | 0.157 (0.021)
  12 Weeks | 0.112 (0.122) | 0.183 (0.067)

9. Secondary Outcome: Change in Serum Glucose
Time Frame: Baseline, 2 weeks, 6 weeks, and 12 weeks
Population: Data no longer exists in the research file depository due it its vintage. Unable to report this measure.
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Other Adverse Events
Description: The Systematic Assessment for Treatment Emergent Events-General Inquiry (SAFTEE-GI) was used to collect and analyze data about potential medication related side effects. Each of 12 subjects was queried using the SAFTEE-GI at 3 time points (1, 2 and 3 weeks) for a possible of 36 adverse event reports.
Time Frame: up to 3 weeks
Measure: Number; unit: incidence of adverse events
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 6 | 6
incidence of adverse events
  Musculoskeletal | 2 | 1
  Sleeplessness | 3 | 0
  Reduced Blood Sugar | 2 | 0
  Decreased Energy | 0 | 1
  Upper Respiratory Infection | 1 | 1
  Increased Mood | 1 | 0
  Mild Urinary Hesitancy | 0 | 1

ADVERSE EVENTS:
Time Frame: up to 3 weeks
Description: There is no longer access to total participants affected by Other Adverse Events, therefore we report 0 participants affected and at risk in this table. Please refer to Outcome Measure 10 where the available Other Adverse Event information for this study is reported.
Arm/Group | Prednisone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes